CLINICAL TRIAL: NCT00664378
Title: A Prospective, Single-arm, Two-stage, Open-label Phase II Trial of CYT997 in Relapsed and Refractory Multiple Myeloma
Brief Title: Efficacy Study of CYT997 in Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty enrolling patients
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCL07001
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2013-04

CONDITIONS: Relapsed and Refractory Multiple Myeloma
Keywords: Multiple myeloma, relapsed, refractory
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — CYT997

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): CYT997
  Interventions: Drug: CYT997

INTERVENTIONS:
Drug: CYT997 — Intravenous infusion (24h); 202mg/m2 on days 1 and 8 of a 21 day cycle

SUMMARY:
This is a clinical research study that is designed to test the safety of CYT997 when given to patients with multiple myeloma and to test if CYT997 has any activity against that cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma per International Working Group (IWG) criteria
* Have received at least 1 but no more than 4 prior lines of therapy
* Have failed to respond to the most recently administered anti-myeloma therapy
* Have a life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status < 3
* At registration absolute neutrophil count > 1x10^9/L and platelet count > 50 x 10^9/L unsupported
* At registration bilirubin less than 1.5 x upper limit of normal and transaminases less than 2 x upper limit of normal and serum creatinine less than 0.19 mmol/L
* Written informed consent
* Must agree to adequate contraceptive measure if indicated

Exclusion Criteria:

* Patients with monoclonal gammopathy of undetermined significance
* Known or suspected hypersensitivity to CYT997
* Patient with uncontrolled intercurrent illness
* Active infections or other illnesses that precludes chemotherapy administration or patient compliance.
* Pregnant or lactating women.
* Patients who have received any other investigational agents in the last 3 weeks prior to the start of treatment.
* Patients with the following conditions will be excluded:

  * myocardial infarction or stroke within 6 months
  * unstable angina pectoris or acute ischemic changes on ECG
  * history of diabetic retinopathy
  * symptomatic peripheral arterial disease
  * major surgery in the last 30 days
* Patients with uncontrolled diarrhea despite optimal medication and those with any history of acute gastrointestinal bleeding
* Patients with a baseline prolongation of the QTc interval of Common Terminology Criteria (CTC) Grade 1 (QTc > 0.45-0.47 sec) or greater
* Patients with impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

  * left ventricular ejection fraction (LVEF) < 45% as determined by multigated acquisition (MUGA) scan or echocardiogram;
  * complete left bundle branch block;
  * obligate use of a cardiac pacemaker;
  * congenital long QT syndrome;
  * history or presence of ventricular tachyarrhythmia;
  * presence of unstable atrial fibrillation (ventricular response > 100 bpm). -Patients with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria;
  * clinically significant resting bradycardia (< 50 bpm);
  * right bundle branch block + left anterior hemiblock (bifascicular block);
  * angina pectoris ≤ 3 months prior to starting study drug;
  * acute myocardial infarction (MI) ≤ 3 months prior to starting study drug; or
  * other clinically significant heart disease (e.g., congestive heart failure (CHF), uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen).
* Patients currently receiving treatment with medications known to prolong the QTc interval and/or to induce Torsades de Pointes arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate to CYT997 when used to treat patients with relapsed or refractory multiple myeloma | Baseline to study completion
  The overall response rate to CYT997 when used to treat patients with relapsed or refractory multiple myeloma once every 3 week cycle

SECONDARY OUTCOMES:
Number of cycles required to achieve maximum response | Baseline to study completion
Overall survival | Baseline to study completion
Safety and tolerability | Baseline to study completion
Time to disease progression | Baseline to study completion

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Spencer, Assoc Prof., Principal Investigator — Myeloma Research Group, The Alfred Hospital, Melbourne
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia